CLINICAL TRIAL: NCT06020144
Title: A Phase 3, Randomized, Double-Blind, Positive-controlled, Head-to-Head Monotherapy Study Comparing TLL-018 to Tofacitinib in Subjects With Active Rheumatoid Arthritis With Inadequate Response or Intolerance to Biologic DMARDs (bDMARDs)
Brief Title: A Phase 3 Study Comparing TLL-018 to Tofacitinib in RA Subjects With Inadequate Response or Intolerance to bDMARDs
Acronym: TARA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLL-018-301
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequence A (Experimental): TLL018 tablets, 2piece,BID
  Interventions: Drug: TLL-018
- sequence B (Active Comparator): Tofacitinib tablets, 1piece,BID
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: TLL-018 — Oral tablets administered 2pieces BID for 52 weeks.
  Other Names: TLL-018 tablets
  Arms: sequence A
Drug: Tofacitinib — Oral tablets administered 1pieces BID for 52 weeks.
  Other Names: Tofacitinib tablets
  Arms: sequence B

SUMMARY:
A randomized, double-blind, double-dummy, positive-controlled, phase 3 study to assess the safety and efficacy of TLL-018 in active rheumatoid arthritis subjects who had an inadequate response or intolerance to Biologic DMARDs.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, tofacitinib-parallel-group, phase 3 study to assess the safety and efficacy of TLL-018 in active rheumatoid arthritis subjects who had an inadequate response or intolerance to Biologic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65;
* Meet the diagnostic criteria of rheumatoid arthritis of the American College of Rheumatology/European Alliance against Rheumatism (ACR/EULAR,2010) with duration of at least 3 months;
* Meet the criteria for active rheumatoid arthritis；
* Have received at least one kind of bDMARDs for three months or longer and show inadequate response or intolerance to at least one kind of bDMARDs；
* Meet the ACR (1991) grading criteria of grade I, II or III；
* Discontinuation of bDMARDs or JAK inhibitors for more than four weeks；
* To sustain a stable status, oral administration of stable doses of glucocorticoids (≤ prednisone 10 mg/day or equivalent corticosteroids) and stable doses of nonsteroidal anti-inflammatory drugs (NSAIDs) are allowed to use, provided that stable doses are maintained for at least one week prior to the study；
* BMI index is less than 35 kg/m2;
* Women of Child Bearing Potential (WOCBP) should not be pregnant or breastfeeding and the pregnancy test should be negative before randomization;
* Subjects (whether male or female) should have adequate barrier contraception during the whole treatment period and at least 90 days after treatment; subjects should avoid the sperm or ovum donation for at least six months after treatment；
* Subjects understand the informed consent form (ICF), volunteer for the study and sign the ICF;

Exclusion Criteria:

* With other rheumatic diseases;
* With other systemic inflammatory diseases;
* With progressive or uncontrolled symptoms of renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiovascular, neurologic, psychiatric, or cerebral disease;
* Previous history of severe hematologic diseases;
* Previous history of malignancy within five years, with exception of cured basal cell carcinoma or cutaneous squamous cell carcinoma or cervical carcinoma in situ.
* With active infection before randomization;
* Herpes zoster occurred within 1 year prior to randomization; disseminated or recurrent herpes zoster prior to randomization; disseminated herpes simplex before randomization;
* Previous history of active tuberculosis (TB) and no evidence of clinical cure or imaging evidence of active TB; or T-spot or PPD positive at screening but have received TB preventive therapy less than one month;
* HBsAg positive (or HBsAg negative but anti-HBc positive and HBV-DNA quantitative test positive), HCV antibody and HCV-RNA positive, or HIV antibody positive;
* Previous history of thrombocytopenia, coagulopathy, or platelet dysfunction;
* Previous history of cardiovascular and cerebrovascular accidents;
* Previous history of thromboembolism or risk factors;
* Previous history of gastrointestinal perforation;
* Temporary usage of NSAIDs within 24 hours prior to the baseline visit;
* Have received anti-rheumatic herb within 4 weeks before randomization;
* Have received interferon therapy within 4 weeks before randomization;
* Have donated blood more than 400 ml or received blood transfusion within 3 months prior to the study;
* Have received any live vaccine within 2 months before randomization or plan to receive a live vaccine during the study;
* Have experienced major surgery within 4 weeks before randomization, or expected to receive major surgical treatment after enrollment;
* Laboratory test results are abnormal and may interfere the study judged by investigators;
* Use of potent opioids within 4 weeks before the baseline visit;
* Allergy to ingredients or excipients of tofacitinib or TLL-018;
* Unable to accomplish evaluation in study;
* Receiving any study drug within 4 weeks or less than 5 elimination of half-life period) before randomization (whichever is longer);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving American College of Rheumatology 50% (ACR50) Response | Week 24
  ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in painful and tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP)at each visit.

SECONDARY OUTCOMES:
Proportion of subjects achieving DAS28-hsCRP <2.6 | Week 24
  Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014*participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity.
Proportion of subjects achieving American College of Rheumatology 20% (ACR20) and 70% (ACR70) Response | Week 24
  ACR20/70 response: greater than or equal to (>=) 20/70 percent (%) improvement in painful and tender joint count; >= 20%/70% improvement in swollen joint count; and >= 20%/70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP)at each visit.
Change From Baseline in Disease Activity Score Based on 28-Joints Count-High-Sensitivity C-reactive Protein (DAS28-hsCRP) | Week 24
  Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014*participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity. Change = value at observation minus value at baseline.
Changes From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score | Week 24
  HAQ-DI score was an evaluation of the functional status for a participant. The 20-question instrument assessed the degree of difficulty a person had in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0, indicated no difficulty, to 3, indicated inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Changes From Baseline in SF-36 Score | Week 24
  SF-36 score was an evaluation of the functional status for a participant,taping eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Coded numeric values are recoded per the scoring key. All items are scored so that a high score defines a more favorable health state. Each item is scored on a o to 100 range. Items in the same scale are averaged together to create the 8 scale scores.
Proportion of subjects achieving DAS28-hsCRP <＝3.2 | Week 24
  Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014*participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity.
Proportion of subjects achieving CDAI <＝10 | Week 24
  Clinical Disease Activity Index equals the sum of score of following variables：Tender joint count (TJC28), Swollen joint count (SJC28), Patient's Global Assessment of Arthritis, Physician's Global Assessment of Arthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No